CLINICAL TRIAL: NCT00000903
Title: A Phase III Randomized, Controlled Trial of Efavirenz (EFV) or Nelfinavir (NFV) in Combination With Fixed-Dose Combination Lamivudine/Zidovudine (3TC/ZDV) and Indinavir (IDV) in HIV-Infected Subjects With Less Than or Equal to 200 CD4 Cells/mm3 or Greater Than or Equal to 80,000 HIV RNA Copies/ml in Plasma
Brief Title: Addition of Efavirenz or Nelfinavir to a Lamivudine/Zidovudine/Indinavir HIV Treatment Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 388; 11347 (Registry Identifier: DAIDS ES); Substudy ACTG 734; Substudy ACTG A5060s; Substudy ACTG 732; Substudy ACTG 733; Substudy ACTG 735; Substudy ACTG 737; Substudy ACTG 746
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Lamivudine; Indinavir; RNA, Viral; Reverse Transcriptase Inhibitors; Nelfinavir; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; lamivudine, zidovudine drug combination; Nelfinavir; efavirenz

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine/Zidovudine
Drug: Nelfinavir mesylate
Drug: Efavirenz

SUMMARY:
To compare time to a virologic failure (first of 2 consecutive plasma HIV RNA levels greater than or equal to 200 copies/ml at or after Week 24) of each 4-drug regimen vs the 3-drug regimen. To determine the safety, tolerance, and virologic benefits of either nelfinavir (NFV) or efavirenz (EFV) with indinavir/lamivudine/zidovudine (IDV/3TC/ZDV) vs IDV/3TC/ZDV alone, in the treatment of patients with advanced HIV disease who have received limited or no prior antiretroviral therapy.

Prior ACTG studies have shown that the 3-drug combination regimen (IDV/ZDV/3TC) resulted in improved clinical outcomes and therefore may prolong the effects of therapy. The enhanced effects seen with combination therapies are likely related to a greater suppression of RNA replication and alterations in resistance patterns. Due to the progressive success of combination regimens, it is possible that more potent regimens will further enhance viral suppression and provide more durable treatment responses. In light of the additive suppression of HIV replication determined by pharmacological, immunological, and virological results, nelfinavir (NFV) as an addition to IDV/ZDV/3TC will be evaluated. Based on the potency of nonnucleoside reverse transcriptase inhibitors (NNRTIs) to suppress viral replication and the effectiveness of 3-drug regimens containing NNRTIs, efavirenz (EFV) will also be evaluated as an addition to IDV/ZDV/3TC.

DETAILED DESCRIPTION:
Prior ACTG studies have shown that the 3-drug combination regimen (IDV/ZDV/3TC) resulted in improved clinical outcomes and therefore may prolong the effects of therapy. The enhanced effects seen with combination therapies are likely related to a greater suppression of RNA replication and alterations in resistance patterns. Due to the progressive success of combination regimens, it is possible that more potent regimens will further enhance viral suppression and provide more durable treatment responses. In light of the additive suppression of HIV replication determined by pharmacological, immunological, and virological results, nelfinavir (NFV) as an addition to IDV/ZDV/3TC will be evaluated. Based on the potency of nonnucleoside reverse transcriptase inhibitors (NNRTIs) to suppress viral replication and the effectiveness of 3-drug regimens containing NNRTIs, efavirenz (EFV) will also be evaluated as an addition to IDV/ZDV/3TC.

Patients with HIV infection, CD4 cell count less than or equal to 200 cells/mm3 or plasma HIV RNA greater than or equal to 100,000 copies/ml, and limited (no prior 3TC, NNRTI, or protease inhibitor) or no prior antiretroviral treatment are randomized to 1 of 3 arms. Patients are stratified by CD4 cell count (less than or equal to 50 cells/mm3 vs greater than 50 cells/mm3), HIV-1 RNA copy number (less than or equal to 40,000 copies/ml vs greater than 40,000 copies/ml), and prior antiretroviral therapy (no therapy vs any therapy), and then randomly assigned to 1 of 3 treatment arms:

Arm 1: 3TC plus ZDV plus IDV. Arm 2: 3TC plus ZDV plus IDV plus EFV. Arm 3: 3TC plus ZDV plus IDV plus NFV. Patients are followed for at least 72 weeks [AS PER AMENDMENT 2/16/99: 96 weeks] beyond the enrollment of the last patient. Patients who experience virologic relapse will have the option of continuing randomized study medications, switching to Step 2 treatment, switching to another ACTG study, or seeking best available therapy for the remaining weeks of the study. Step 2 treatment consists of abacavir or 2 NNRTIs plus efavirenz plus amprenavir or another protease inhibitor. [AS PER AMENDMENT 4/3/00: Optimally, Step 2 treatment regimens should contain 3 or 4 drugs to which the virus is susceptible. If this is not possible, a drug to which the virus is partially susceptible is acceptable, but a drug to which the virus is resistant should not be included.]

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chemoprophylaxis for Pneumocystis carinii pneumonia.
* Topical and oral antifungal agents (except for oral ketoconazole and itraconazole).
* All antibiotics as clinically indicated (unless otherwise excluded).
* Treatment, maintenance, or chemoprophylaxis with approved agents for opportunistic infections as clinically indicated (unless otherwise excluded).
* Systemic corticosteroids for 21 days or less for acute problems.
* Recombinant erythropoietin (rEPO) and granulocyte colony-stimulating factor (G-CSF, filgrastim).
* Regularly prescribed medications such as antipyretics, analgesics, allergy medications, antidepressants, sleep medications, oral contraceptives, megestrol acetate, testosterone.
* Alternative therapies such as vitamins. Patients should report the use of these therapies.
* [AS PER AMENDMENT 2/16/99: Rifabutin can be administered at a reduced dose.]
* [AS PER AMENDMENT 4/3/00: Systemic cytotoxic chemotherapy. Study team should be notified.]
* [AS PER AMENDMENT 4/3/00: Expanded access and compassionate use drugs are allowed as part of Step 2 treatment only.]

Allowed with caution:

* [AS PER AMENDMENT 4/3/00: Viagra (sildenafil citrate) at a reduced dose unless otherwise approved by the protocol chair.]
* [AS PER AMENDMENT 4/3/00: Lovastatin or simvastatin with PIs is not recommended. Caution should be exercised with the use of all other statins when used concomitantly with PIs.]

Concurrent Treatment:

Allowed:

* Alternative therapies such as acupuncture and visualization techniques. Patients should report use of these therapies.

Patients must have:

* Documented HIV-1 infection.
* CD4 count less than or equal to 200 cells/mm3 or a plasma HIV RNA greater than or equal to 100,000 copies/ml [AS PER AMENDMENT 2/16/99:
* 80,000 copies/ml] within 60 days prior to entry.
* Other lab values performed within 14 days prior to entry.

Prior Medication:

Allowed:

* Zidovudine (ZDV), didanosine (ddI), stavudine (d4T), or zalcitabine (ddC) therapy alone or in combination any time prior to study entry.

Exclusion Criteria

Concurrent Medication:

Excluded:

* All antiretroviral therapies other than study medications. [AS PER AMENDMENT 4/3/00: Compassionate use and expanded access drugs are allowed as part of Step 2 treatment.]
* Investigational drugs without specific approval from the Study Chair. [AS PER AMENDMENT 4/3/00: Compassionate use and expanded access drugs are allowed as part of Step 2 treatment.]
* Systemic cytotoxic chemotherapy. [AS PER AMENDMENT 4/3/00: Systemic cytotoxic chemotherapy is allowed. Study team should be notified.]
* Alprazolam, amiodarone, astemizole, bepridil, bupropion, cisapride, clorazepate, clozapine, diazepam, encainide, ergot alkaloids and derivatives of ergot alkaloids, estazolam, flecainide, flurazepam, itraconazole , ketoconazole, meperidine, midazolam, piroxicam, propafenone, propoxyphene, quinidine, rifabutin, rifampin, terfenadine, triazolam, or zolpidem. [AS PER AMENDMENT 2/16/99: Amiodarone, astemizole, cisapride, ergot alkaloids or drugs containing derivatives of ergot alkaloids, itraconazole, midazolam, triazolam, quinidine, rifampin, terfenadine.] [AS PER AMENDMENT 4/3/00: Amiodarone, astemizole, bepridil, cisapride, ergot alkaloids and derivatives of ergot alkaloids, Hypericum perforatum (St. John's wort), itraconazole, midazolam, quinidine, rifampin, terfenadine, triazolam.]
* Vitamin E supplements. [AS PER AMENDMENT 4/3/00: Multivitamins containing vitamin E are allowed.]

Avoided:

* Herbal medications. Patients should report use.

Patients with the following prior conditions are excluded:

* Acute therapy for an infection or other medical illnesses within 14 days prior to study entry. [AS PER AMENDMENT 2/16/99: Acute therapy for a serious infection or other serious medical illnesses that are potentially life-threatening and require systemic therapy and/or hospitalization within 14 days of study entry.]

Prior Medication:

Excluded within 30 days prior to entry:

* More than 1 day experience with lamivudine (3TC), nonnucleoside reverse transcriptase inhibitor, or protease inhibitor.
* Erythropoietin, G-CSF, or GM-CSF.
* Interferons, interleukins, HIV vaccines, or any experimental therapy.

Excluded within 14 days prior to entry:

* Alprazolam (Xanax), amiodarone (Cordarone), astemizole (Hismanal), bepridil (Vascor), bupropion (Wellbutrin, Zyban), cisapride (Propulsid), clorazepate (Tranxene), clozapine (Clozaril), diazepam (Valium), encainide (Enkaid), ergot alkaloids or drugs containing derivatives of ergot alkaloids, estazolam (ProSom), flecainide (Tambocor), flurazepam (Dalmane), itraconazole (Sporanox), ketoconazole (Nizoral), meperidine (Demerol), midazolam (Versed), piroxicam (Feldene), propafenone (Rythmol), propoxyphene (Darvon, Darvocet), quinidine, rifabutin (Mycobutin), rifampin (Rifadin, Rifamate, Rifater, Rimactane), terfenadine (Seldane), triazolam (Halcion), or zolpidem (Ambien). [AS PER AMENDMENT 2/16/99: Agents excluded within 14 days prior to entry are now as follows:
* amiodarone, astemizole, cisapride, ergot alkaloids or drugs containing derivatives of ergot alkaloids, itraconazole, midazolam, quinidine, rifampin, terfenadine, and triazolam.

Note:

* Rifabutin can be administered at a reduced dose of 150 mg/day.]

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 444
Dates: Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Fischl, Study Chair; Ann Collier, Study Chair; Judith Feinberg, Study Chair; Stefano Vella, Study Chair
Locations (50):
- United States (49):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Marin County Dept. of Health & Human Services, HIV/AIDS Program & Specialty Clinic, San Rafael, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Howard University Hosp., Div. of Infectious Diseases, ACTU, Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS, Miami, Florida
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Weiss Memorial Hosp., Chicago, Illinois
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - Cornell CRS, New York, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - Cornell University A2201, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Weill Med. College of Cornell Univ., The Cornell CTU, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Carolinas Med. Ctr., Charlotte, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico

REFERENCES:
- [Result] Fischl MA, Ribaudo HJ, Collier AC, Erice A, Giuliano M, Dehlinger M, Eron JJ Jr, Saag MS, Hammer SM, Vella S, Morse GD, Feinberg JE, Demeter LM, Eshleman SH; Adult AIDS Clinical Trials Group 388 Study Team. A randomized trial of 2 different 4-drug antiretroviral regimens versus a 3-drug regimen, in advanced human immunodeficiency virus disease. J Infect Dis. 2003 Sep 1;188(5):625-34. doi: 10.1086/377311. Epub 2003 Aug 15. PMID 12934177
- [Result] Demeter LM, Ribaudo HJ, Erice A, Eshleman SH, Hammer SM, Hellmann NS, Fischl MA; AIDS Clinical Trials Group Protocol 388. HIV-1 drug resistance in subjects with advanced HIV-1 infection in whom antiretroviral combination therapy is failing: a substudy of AIDS Clinical Trials Group Protocol 388. Clin Infect Dis. 2004 Aug 15;39(4):552-8. doi: 10.1086/422518. Epub 2004 Jul 30. PMID 15356820
- [Result] DiCenzo R, Forrest A, Fischl MA, Collier A, Feinberg J, Ribaudo H, DiFrancecso R, Morse GD; AIDS Clinical Trials Group 388/733/5060 Study Team. Pharmacokinetics of indinavir and nelfinavir in treatment-naive, human immunodeficiency virus-infected subjects. Antimicrob Agents Chemother. 2004 Mar;48(3):918-23. doi: 10.1128/AAC.48.3.918-923.2004. PMID 14982784
- [Derived] Lok JJ, Hunt PW, Collier AC, Benson CA, Witt MD, Luque AE, Deeks SG, Bosch RJ. The impact of age on the prognostic capacity of CD8+ T-cell activation during suppressive antiretroviral therapy. AIDS. 2013 Aug 24;27(13):2101-10. doi: 10.1097/QAD.0b013e32836191b1. PMID 24326304